CLINICAL TRIAL: NCT04135430
Title: Parental Assessment of the Quality of Life of Infants Under 12 Months of Age With Moderate Bronchiolitis Referred for Ambulatory Respiratory Physiotherapy
Brief Title: Parental Assessment of the Quality of Life of Infants With Bronchiolitis Episodes
Acronym: BRONKILIB3
Status: Completed | Type: Observational
Sponsor: Association des Réseaux Bronchiolite (Unknown)
Responsible Party: Sponsor
Other Study IDs: BRONKILIB3; 2019-A01633-54 (Other: ID-RCB)
Record Dates: First submitted 2019-09-30; First posted 2019-10-22 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Infants; Chest physiotherapy
MeSH Terms: conditions — Bronchiolitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: Practice of an updated questionnaire at D0, D2 and D7
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — practice of an updated questionnaire at D0, D2 and D7

SUMMARY:
Infant bronchiolitis is a frequent pathology that is the cause of a very large number of medical outpatient and physiotherapy treatments in France. Many international studies and recommendations have invalidated any drug treatment during its management during the first episode. In France, the consensus conference promoted by the National Agency for Accreditation and Health Evaluation (ANAES) in September 2000 was in the same vein.

Regarding the respiratory physiotherapy component, posture drainage, vibration and percussion are not considered effective. ANAES recommended the use of respiratory physiotherapy with passive exhalation techniques. This is a method of care that has developed mainly in French-speaking countries, making it difficult to compare with the habits of Anglo-Saxon countries, which, more generally, do not prescribe it. In France, the level of evidence of its effectiveness is considered low (grade C). To date, the vast majority of studies have focused exclusively on a population of infants hospitalized for severe bronchiolitis. For this type of population, the value of such treatment to shorten the healing time has not been demonstrated. So much so that the ANAES, in its time, recommended that studies be carried out "on an outpatient basis" to assess their degree. In this respect, several recent studies have provided new data. Despite the reservations inherent in their methodologies and/or staff, they raise the question of the interest of the respiratory physiotherapy on an outpatient basis. In terms of professional practice, the American recommendations state that clinicians should educate family members about evidence-based diagnosis, treatment and prevention in bronchiolitis. Finally, an opinion survey concludes that holders of parental authority are seeking information on bronchiolitis and that approximately 90% have read the brochure given out of the maternity ward explaining the modes of transmission, manifestations, care and hygiene measures in the event of bronchiolitis. Pending new French recommendations, it seems legitimate to evaluate the level of perception of the effect of pediatric respiratory physiotherapy with increase in expiratory flow (IEF) in urban practice on the respiratory comfort of infants directly with families confronted with this pathology.

DETAILED DESCRIPTION:
Infant bronchiolitis is a frequent pathology that is the cause of a very large number of medical outpatient and physiotherapy treatments in France. Many international studies and recommendations have invalidated any drug treatment during its management during the first episode. In France, the consensus conference promoted by the National Agency for Accreditation and Health Evaluation (ANAES) in September 2000 was in the same vein.

Regarding the respiratory physiotherapy component, posture drainage, vibration and percussion are not considered effective. ANAES recommended the use of respiratory physiotherapy with passive exhalation techniques. This is a method of care that has developed mainly in French-speaking countries, making it difficult to compare with the habits of Anglo-Saxon countries, which, more generally, do not prescribe it. In France, the level of evidence of its effectiveness is considered low (grade C). To date, the vast majority of studies have focused exclusively on a population of infants hospitalized for severe bronchiolitis. For this type of population, the value of such treatment to shorten the healing time has not been demonstrated. So much so that the ANAES, in its time, recommended that studies be carried out "on an outpatient basis" to assess their degree. In this respect, several recent studies have provided new data. Despite the reservations inherent in their methodologies and/or staff, they raise the question of the interest of respiratory physiotherapy in ambulatory care. In terms of professional practice, the American recommendations state that clinicians should educate family members about evidence-based diagnosis, treatment and prevention in bronchiolitis. Finally, an opinion survey concludes that holders of parental authority are seeking information on bronchiolitis and that approximately 90% have read the brochure given out of the maternity ward explaining the modes of transmission, manifestations, care and hygiene measures in the event of bronchiolitis. Pending new French recommendations, it seems legitimate to evaluate the level of perception of the effect of pediatric respiratory physiotherapy with increase in expiratory flow (IEF) in urban practice on the respiratory comfort of infants directly with families confronted with this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Infant up to 12 months of age
* Wang's score ≥ at 4 and < 9
* With first or second episode of bronchiolitis with a medical prescription for respiratory physiotherapy in the city.
* Consultation for a first session, or second session of respiratory physiotherapy

Exclusion Criteria:

* History or atopic predisposition
* History(s) of prematurity (34 weeks of amenorrhea or less)
* History of bronchopulmonary dysplasia
* Underlying heart disease, severe chronic lung disease
* Contraindication to the use of Kinesitherapy: prolonged corticosteroid therapy (more than one month), rickets, osteogenesis imperfecta, thrombocytopenia, rib fracture
* Opposition of holders of parental authority

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants up to 12 months of age with first or second episode bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-04-04 (Actual)

PRIMARY OUTCOMES:
QUALIN score | 24 hours
  Evolution of the Quality of life of infants and young children (QUALIN) score between before the session and 12 to 24 hours after the session.

SECONDARY OUTCOMES:
Questionnaire about accessibility of the care chain | 8 days
  This is a questionnaire that has not been validated in the literature. Its purpose is to assess the feelings of holders of parental authority about the conditions of access to outpatient care.
Questionnaire about understanding of the information | 8 days
  This is a questionnaire that has not been validated in the literature. The purpose of this questionnaire is to evaluate the parent's feelings about understanding information
Questionnaire about perceived professional competence. | 8 days
  This is a questionnaire that has not been validated in the literature. The purpose of this questionnaire is to evaluate the parent's feelings about perceived professional competence
Questionnaire about security of care | 8 days
  This is a questionnaire that has not been validated in the literature. The purpose of this questionnaire is to evaluate the parent's feelings about perceived professional competence The security of care
Questionnaire about child's respiratory comfort | 8 days
  This is a questionnaire that has not been validated in the literature. The purpose of this questionnaire is to evaluate the parent's feelings about the evolution of their child's respiratory comfort after the physiotherapy session.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Rb Picard, Amiens
  - RB 74, Annecy-le-Vieux
  - GAB, Arpajon
  - Aquirespi, Bordeaux
  - Rb Loiret, Fleury-les-Aubrais
  - La Rochelle, La Rochelle
  - Occirespi, Léguevin
  - Rb Grand Est, Malzéville
  - ARBAM, Marseille
  - CHU Robert-Debré, Paris
  - RB 59 62, Seclin

IPD SHARING:
Plan to Share IPD: No